CLINICAL TRIAL: NCT05270187
Title: Efficacy of Multiwave Locked System Laser on Recovery of Patients With Bell's Palsy: A Randomized Placebo Controlled Trial.
Brief Title: Multiwave Locked System Laser for Patients With Bell's Palsy.
Acronym: MLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Mohamed Alayat, Associate Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-MED-10023150
Record Dates: First submitted 2022-01-19; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Facial Paralyses, Idiopathic; Laser Therapy; Bell Palsy
Keywords: Bell's palsy; Multiwave locked system laser therapy; facial disability scale; House-Brackmann scale
MeSH Terms: conditions — Bell Palsy | interventions — Low-Level Light Therapy; Laser Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: A total of 60 recruited patients will be randomly assigned into three groups of 20 patients in each. Group one will receive MLS laser therapy with 10 J/cm2 in scanning mode to the affected side plus facial massage and exercises. Group two will receive MLS laser therapy to predetermined eight motor points to facial muscles plus facial massage and exercises. Group three will receive placebo laser plus facial massage and exercises.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: By sealed envelopes, the allocation concealment will be achieved. Patient randomization is performed simply by computer number generator for each patient using GraphPad software. All eligible participants will be evaluated by independent physician and will be treated by the same therapist. The physician conducts the processes of participant enrollment, and allocation. The same assessors will measure the measured outcome. Both the therapist and the assessor will be blinded (masked) from patient's enrollment into the three study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scanning Gorup (Experimental): Patients in this group will receive facial massage, facial expression exercises and a Multiwave Locked System Laser with energy density 10 J/cm2. Laser will scan the affected side after calculating the distance and the total energy delivered to the one side of the face.
  The average treatment area is 50 cm2. The energy density was 10 J/cm2 with a total energy of 500 J and the treatment time is approximately 15 minutes. The laser probe will be away from the eye region. Both patients and therapist wear a laser googles.
  Interventions: Other: Photobiomodulation therapy (laser therapy); Other: Facial massage and facial expression exercises
- Point laser Group (Experimental): Patients in this group will received facial massage, facial expression exercises and laser at predetermined eight points on the affected side of the facial muscles. the hand piece is positioned perpendicular to 8 points which is located on the superficial roots of the facial nerve of the affected side. Each point will receive an energy density of 10 J/point with total energy delivered to the patient during one session of 80 joules. The time of application 90 sec/point. laser is calibrated by the manufacture company before the starting the experiment and periodically during the sessions. The laser probe will be away from the eye region. Both patients and therapist wear a laser googles.
  Interventions: Other: Photobiomodulation therapy (laser therapy); Other: Facial massage and facial expression exercises
- Control Group (Placebo Comparator): patients in this group will receive only facial massage, facial expression exercises and placebo laser. Facial expression exercises include active graduated strengthening exercises in front of a mirror (active assisted, freedom, and resisted), proprioceptive neuromuscular facilitation exercises for facial muscles, and resisted exercises for neck muscles. Participants are taught to perform massage and exercises correctly by the physiotherapist. All treatment groups are given instruction to repeat the massage and exercises two times a day for at least 6 weeks. The patient or one of his/her family members will confirm that the participant carries out the massage and exercises at home.
  Interventions: Other: Facial massage and facial expression exercises

INTERVENTIONS:
Other: Photobiomodulation therapy (laser therapy) — The Multiwave Locked System Laser will treat both the scan and point application groups. M6 laser equipment (ASA, Arcugnano, Italy) is used in this study in the physiotherapy and rehabilitation department, Faculty of Applied Medical Science, Umm Al-Qura University. It provides synchronized and overlapping continuous and pulsed emissions of Ga-Al-Ar laser emitted in a single hand piece. M6 has a continuous emission of a wavelength of 808 nm with peak power of 1000 mW, mean power of 500mW, spot diameter of 2 cm, and spot area of 3.14 cm2. Pulsed emission has a wavelength of 905 nm, peak power of 25 W, and mean power of 54mW with frequency of 1500 Hz.
  Other Names: Multiwave Locked System Laser
  Arms: Point laser Group; Scanning Gorup
Other: Facial massage and facial expression exercises — Facial massage and facial expression exercises will be applied for all patients in the three treatment groups. It includes simple facial expression exercises, active graduated strengthening exercises in front of a mirror (active assisted, freedom, and resisted), proprioceptive neuromuscular facilitation exercises for facial muscles, and resisted exercises for neck muscles. Participants are taught to perform massage and exercises correctly by the physiotherapist. All treatment groups are given instruction to repeat the massage and exercises two times a day for at least 6 weeks. The patient or one of his/her family members will confirm that the participant carries out the massage and exercises at home.
  Other Names: Exercises

SUMMARY:
Background: Idiopathic Bell's palsy (IBP) is a unilateral facial paralysis of sudden onset and unknown etiology. Patient with IBP has an impaired facial expressions and psychological affection, which interfere with social communication. Multiwave locked system (MLS) laser therapy is a class IV laser with synchronizes emission of an 808 nm continuous laser and a 905 nm pulsed laser. It is proposed that MLS facilitates greater penetration and therapeutic effects than low-level laser therapy (LLLT).

Aims: The aim of present study is to investigate the effect of MLS laser in the treatment of patients with unilateral IBP.

Participant: A total number of 60 patients with IBP will be recruited from Makkah hospitals. Treatment will begin in the subacute phase as they referred from neuro-doctors. All the recruited patients will be randomly assigned into three groups of 20 patients each.

Intervention: All patients will be treated with facial massage and exercises. In addition, group one will receive MLS laser with 10 J/cm2 in scanning mode while the group two will receive 10J/point for eight points.

Measured variables: Facial disability scale (FDI) and House-Brackmann scale HBS will used to assess the grade of facial nerve recovery. The scores of both questionnaires will be collected at the baseline, after three and six weeks after treatment.

Statistical Analysis: The Friedman and Wilcoxon signed ranks tests will be used to compare the FDI and HBS scores within each group

DETAILED DESCRIPTION:
Multi-wave locked system (MLS) laser therapy had been presented in the arena of rehabilitation and attained interests of numerous researchers due to its unique features. MLS laser is a Class IV, high-power laser, which is characterized by a combination of two waveforms of continuous emissions of an 808 nm wavelength and a pulsed 905 nm emitted in synchrony. MLS used recently in research and revealed significant reduction of musculoskeletal pain and disability. Researchers recommend its use in case of muscle lesions and/or diseases. No proved way was shown to use laser in the treatment of facial palsy in either scanning the affected side or applying laser to specific motor points.

It was proposed that the combination of the dual laser waveforms offers better penetrability and outcomes on than ordinary lasers and help in recovery of facial muscle.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has unilateral IBP either on the right or left side.
* Treatment will begin in the sub-acute stage of illness 3-5 days after the acute onset subsided.
* patients will accept to attend to the physical therapy department to receive their corresponding treatment twice a week for successive six weeks.

Exclusion Criteria:

* Patients who have central nervous system pathology
* sensory loss over the face, or recurrence of BP.
* Patients with upper motor facial nerve palsy will be also excluded.
* Any infant or child (≤18 years) with BP will be also excluded.
* Chronic facial palsy patients
* Patients BP having after a tumor, stroke, and Lyme disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Facial disability scale (FDI) | The scores of the questionnaire will be collected at the baseline before treatment.
  The FDI was produced by Van Swearingen and Brach to improve the assessment of facial neuromuscular dysfunction. Beyond the impairment domain, this index provides a reliable measurement with construct validity for evaluating patients with facial nerve disorders.
Facial disability scale (FDI) | The scores of the questionnaire will be collected after three weeks after treatment.
  The FDI was produced by Van Swearingen and Brach to improve the assessment of facial neuromuscular dysfunction. Beyond the impairment domain, this index provides a reliable measurement with construct validity for evaluating patients with facial nerve disorders.
Facial disability scale (FDI) | The scores of the questionnaire will be collected after six weeks after treatment.
  The FDI was produced by Van Swearingen and Brach to improve the assessment of facial neuromuscular dysfunction. Beyond the impairment domain, this index provides a reliable measurement with construct validity for evaluating patients with facial nerve disorders.

SECONDARY OUTCOMES:
House-Brackmann scale (HBS) | The scores of the questionnaire will be collected at the baseline before starting of the treatment
  This scale analyses the symmetry, synkinesis, stiffness, and global mobility of the face [6]. It consists of six divisions (normal, mild dysfunction, moderate dysfunction, moderately severe dysfunction, severe dysfunction, and total paralysis) with grade one indicating a normal facial function in all areas and grade six indicating total paralysis.
House-Brackmann scale HBS | The scores of the questionnaire will be collected after three weeks after treatment.
  This scale analyses the symmetry, synkinesis, stiffness, and global mobility of the face [6]. It consists of six divisions (normal, mild dysfunction, moderate dysfunction, moderately severe dysfunction, severe dysfunction, and total paralysis) with grade one indicating a normal facial function in all areas and grade six indicating total paralysis.
House-Brackmann scale HBS | The scores of the questionnaire will be collected after six weeks after treatment.
  This scale analyses the symmetry, synkinesis, stiffness, and global mobility of the face [6]. It consists of six divisions (normal, mild dysfunction, moderate dysfunction, moderately severe dysfunction, severe dysfunction, and total paralysis) with grade one indicating a normal facial function in all areas and grade six indicating total paralysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alayat, Principal Investigator — Associate Professor of Physical Therapy, Faculty of Applied Medical Science
Locations (1):
- Umm Al-Qura University, Faculty of Applied Medical Science, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alayat MS, Elsodany AM, El Fiky AA. Efficacy of high and low level laser therapy in the treatment of Bell's palsy: a randomized double blind placebo-controlled trial. Lasers Med Sci. 2014 Jan;29(1):335-42. doi: 10.1007/s10103-013-1352-z. Epub 2013 May 26. PMID 23709010
- [Result] Alayat MS, Elsoudany AM, Ali ME. Efficacy of Multiwave Locked System Laser on Pain and Function in Patients with Chronic Neck Pain: A Randomized Placebo-Controlled Trial. Photomed Laser Surg. 2017 Aug;35(8):450-455. doi: 10.1089/pho.2017.4292. PMID 28783464
- [Result] Shafshak TS. The treatment of facial palsy from the point of view of physical and rehabilitation medicine. Eura Medicophys. 2006 Mar;42(1):41-7. PMID 16565685
- [Result] VanSwearingen JM, Brach JS. The Facial Disability Index: reliability and validity of a disability assessment instrument for disorders of the facial neuromuscular system. Phys Ther. 1996 Dec;76(12):1288-98; discussion 1298-300. doi: 10.1093/ptj/76.12.1288. PMID 8959998
- [Result] Yen TL, Driscoll CL, Lalwani AK. Significance of House-Brackmann facial nerve grading global score in the setting of differential facial nerve function. Otol Neurotol. 2003 Jan;24(1):118-22. doi: 10.1097/00129492-200301000-00023. PMID 12544040
- [Result] Lindsay RW, Robinson M, Hadlock TA. Comprehensive facial rehabilitation improves function in people with facial paralysis: a 5-year experience at the Massachusetts Eye and Ear Infirmary. Phys Ther. 2010 Mar;90(3):391-7. doi: 10.2522/ptj.20090176. Epub 2010 Jan 21. PMID 20093325